CLINICAL TRIAL: NCT02169024
Title: Development of a Nationally Scalable Model of Group Prenatal Care to Improve Birth Outcomes: "Expect With Me"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: United Health Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1304011772
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Pregnancy; Premature Birth; Infant, Low Birth Weight; Postpartum Period; Sexually Transmitted Diseases
Keywords: prenatal care; group care; Expect With Me; evaluation studies; group prenatal care
MeSH Terms: conditions — Premature Birth; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Expect With Me group prenatal care vs. Individual Care Only prenatal care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expect With Me group prenatal care (Experimental): receiving prenatal care through an Expect With Me group
  Interventions: Behavioral: Expect With Me group prenatal care
- Individual Care Only (Active Comparator): Standard of Care- individual prenatal care
  Interventions: Other: Standard individual prenatal care

INTERVENTIONS:
Behavioral: Expect With Me group prenatal care — Expect With Me group prenatal care was designed based on: principles of group care; evidence from RCTs demonstrating improved birth outcomes; ACOG clinical guidelines; and research on patient and provider engagement through technology. Designed with national dissemination as a primary consideration, Expect With Me incorporates best evidence-based aspects of existing models of group care, with a novel IT platform to improve patient engagement and support, enhance health behaviors and decision making, connect providers and patients, and improve health service delivery. Expect With Me provides care to groups of 8-12 women of the same gestational age, implemented after initial individual assessment through delivery. Group visits are 90-120 minutes each, and follow a structured curriculum that incorporates standard content of prenatal care, and emphasizes critical health issues relevant to pregnancy, such as nutrition, physical activity, stress/mental health and sexual health.
  Other Names: group prenatal care
  Arms: Expect With Me group prenatal care
Other: Standard individual prenatal care — Standard of care- individual prenatal care
  Other Names: Individual Care Only
  Arms: Individual Care Only

SUMMARY:
This study addresses the intractable challenges of adverse birth outcomes, including preterm delivery and low birthweight, by proposing the development, implementation and evaluation of a model of group prenatal care that could be scaled nationally. Group prenatal care models have been demonstrated through rigorous research to provide significantly improved birth outcomes with implications for maternal-child health and substantial cost savings. However, group prenatal care is currently available to only a small fraction of the more than four million women who give birth annually in the US. Through the development, implementation and evaluation of a new model of group prenatal care, we will create an outcomes-focused model of group prenatal care that will be scalable nationally with an eye toward improving US birth outcomes.

The long-term objective of the proposed study is to reduce the risk for adverse perinatal outcomes during and after pregnancy among women and families receiving prenatal care in health centers in 3 geographic locations serving vulnerable populations: Hidalgo County Texas, Nashville Tennessee, and Detroit Michigan. We will develop, disseminate, and evaluate a new and improved model of group prenatal care, "Expect with Me," based on our previous research on group models of prenatal care, which has already yielded favorable behavioral and biological results in two randomized controlled trials.

We hypothesize that, relative to women who receive standard individual prenatal care, the women who receive "Expect with Me" group prenatal care will be significantly more likely to:

1. have better perinatal outcomes, including better health behaviors during pregnancy (e.g., nutrition, physical activity), better birth outcomes (e.g., decreased preterm labor, low birthweight, Neonatal Intensive Care Unit stays), and better postpartum indicators (e.g., increased breastfeeding);
2. report greater change in risk-related behaviors and psychosocial characteristics that could be considered potential mechanisms for the program's effectiveness;
3. have lower rates of sexually transmitted diseases and rapid repeat pregnancy one year postpartum;
4. have lower healthcare costs through improved outcomes (e.g., appropriate care utilization, fewer complications, reduced NICU admissions/length of stays)

Comparisons based on propensity-score matched sample of women receiving standard individual prenatal care at the same clinical sites.

DETAILED DESCRIPTION:
This study addresses the intractable challenges of adverse birth outcomes, including preterm delivery and low birthweight, by proposing the development, implementation and evaluation of a model of group prenatal care that could be scaled nationally. Group prenatal care models have been demonstrated through rigorous research to provide significantly improved birth outcomes with implications for maternal-child health and substantial cost savings. However, group prenatal care is currently available to only a small fraction of the more than four million women who give birth annually in the US. Through the development, implementation and evaluation of a new model of group prenatal care, we will create an outcomes-focused model of group prenatal care that will be scalable nationally with an eye toward improving US birth outcomes.

Specific Aims:

The long-term objective of the proposed study is to reduce the risk for adverse perinatal outcomes during and after pregnancy among women and families receiving prenatal care in health centers in 3 geographic locations serving vulnerable populations: Hidalgo County Texas, Nashville Tennessee, and Detroit Michigan. We will develop, disseminate, and evaluate a new and improved model of group prenatal care, "Expect with Me," based on our previous research on group models of prenatal care, which has already yielded favorable behavioral and biological results in two randomized controlled trials. The overall objective of this project is to improve maternal health and reduce adverse birth outcomes. We will meet this objective by achieving three specific goals:

1. Develop a new and improved model of group prenatal care, including curriculum, training materials, IT infrastructure and marketing materials to support broad adoption of group prenatal care, enhance consumer experience, monitor patient outcomes, and ensure national scalability.
2. Implement group prenatal care in three communities at high risk for adverse perinatal outcomes (Hidalgo County TX, Nashville TN, Detroit MI), engaging and training providers in group facilitation and the established curriculum, engaging patients through improved in-reach and outreach strategies, and implementing IT infrastructure to improve uptake, patient experience, and sustainability through the monitoring of patient outcomes.
3. Evaluate the effect of implementing group prenatal care through a rigorous process and outcome evaluation that identifies any barriers to national scalability and examines maternal health and birth outcomes and resultant cost implications.

Specific Study Hypotheses

We hypothesize that, relative to women who receive standard individual prenatal care, the women who receive "Expect with Me" group prenatal care will be significantly more likely to:

1. have better perinatal outcomes, including better health behaviors during pregnancy (e.g., nutrition, physical activity), better birth outcomes (e.g., decreased preterm labor, low birthweight, Neonatal Intensive Care Unit stays), and better postpartum indicators (e.g., increased breastfeeding);
2. report greater change in risk-related behaviors and psychosocial characteristics that could be considered potential mechanisms for the program's effectiveness;
3. have lower rates of sexually transmitted diseases and rapid repeat pregnancy one year postpartum;
4. have lower healthcare costs through improved outcomes (e.g., appropriate care utilization, fewer complications, reduced NICU admissions/length of stays)

ELIGIBILITY:
Inclusion Criteria:

* less than 24 weeks pregnant
* able to attend groups conducted in English or Spanish
* consent to share their data with the study

Exclusion Criteria:

* severe medical problem requiring individual care only, as determined by the participating clinical practice

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2402 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Risk of preterm birth incidence | up to 37 weeks gestation
  Incidence risk of delivery before 37 weeks gestation
Risk of low birth weight incidence | delivery
  Incidence risk of infant weight at birth < 2500 grams
Risk of small for gestational age incidence | delivery
  Incidence risk of infant weight below the 10th percentile for the gestational age at birth
Risk of neonatal intensive care unit (NICU) admission incidence | birth
  Incidence risk of being admitted to the neonatal intensive care unit (NICU) at birth

SECONDARY OUTCOMES:
breastfeeding | 6 and 12 months postpartum
  initiation and duration of breastfeeding
nutrition | 2nd and 3rd trimester of pregnancy and 6 and 12 months postpartum
  nutritional choices, food security, and use of mindful eating practices
physical activity | 2nd and 3rd trimester and 6 and 12 months postpartum
  level of physical activity in a typical week
readiness for labor and delivery | measured at 2nd and third trimester
  readiness for labor and delivery
readiness for taking care of baby | 2nd and 3rd trimester of pregnancy
  readiness for taking care of baby
social support | 2nd and 3rd trimester and 6 and 12 months postpartum
  multidimensional scale of perceived social support subscale
condom use self-efficacy | 2nd and 3rd trimester and 6 and 12 months postpartum
  condom use self efficacy scale
substance use | 2nd and 3rd trimester and 6 and 12 months postpartum
  use of cigarettes, alcohol, and drugs
care satisfaction | 3rd trimester
  satisfaction with Expect With Me group prenatal care and use of program components
adherence to medical recommendations | 6 & 12 months postpartum
  adherence to medical recommendations (e.g., 6-week postpartum check, pediatric visits, vaccinations, infant feeding)
postpartum body mass index | measured at 6 and 12 months postpartum
  individual's body weight divided by the square of their height (kg/m2)
maternal weight gain | measured at 2nd and 3rd trimester and birth
  weight gain as compared to medical recommendations
mode of delivery | delivery
  mode of delivery (e.g., cesarean, vaginal)
sexual risk: condom use | measured at 2nd and 3rd trimester and 6 and 12 months postpartum
  condom use percent (0-100%)
sexual risk: contraceptive use (LARC) | measured at 2nd and 3rd trimester and 6 and 12 months postpartum
  use of other contraceptives to prevent pregnancy (no/yes)
sexual risk: number of sexual partners | measured at 2nd and 3rd trimester and 6 and 12 months postpartum
  number of partners
sexual risk: sexually transmitted infection | measured at 2nd and 3rd trimester and 6 and 12 months postpartum
  sexually transmitted infection (no/yes, during pregnancy or incident postpartum)

OTHER OUTCOMES:
nurse visitation | 2nd and 3rd trimester of pregnancy
  participation in a nurse visitation program
sexual debut | 2nd trimester pregnancy
  age at first intercourse
living situation | 2nd and 3rd trimester and 6 and 12 months postpartum
  where and with whom they live with and the stability of their housing
transfer of motivation | 2nd and3rd trimester and 6 and 12 months postpartum
  relation of motivation for self and baby's health
confidence in parenting skills | 6 and 12 months postpartum
  confidence in parenting skills
intimate partner violence | measured at 2nd and 3rd trimester and 6 and 12 months postpartum
  perpetration and victimization of violence by an intimate partner
perceived stress | 2nd and 3rd trimester and 6 and 12 months postpartum
  stress level as reported by patient
depressive symptomatology | 2nd and 3rd trimester of pregnancy
  patient endorsement of depressive symptoms
perceived discrimination | 2nd and 3rd trimester of pregnancy and 6 and 12 months postpartum
  patient experiences of discrimination
resilience | 2nd and 3rd trimester of pregnancy and 6 and 12 months postpartum
  shift and persist scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeannette R Ickovics, Ph.D., Principal Investigator — Yale School of Public Health; Jessica B Lewis, PhD, MFT, Study Director — Yale School of Public Health
Locations (2):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masters C, Carandang RR, Lewis JB, Hagaman A, Metrick R, Ickovics JR, Cunningham SD. Group prenatal care successes, challenges, and frameworks for scaling up: a case study in adopting health care innovations. Implement Sci Commun. 2024 Mar 4;5(1):20. doi: 10.1186/s43058-024-00556-1. PMID 38439113
- [Derived] Lewis JB, Cunningham SD, Shabanova V, Hassan SS, Magriples U, Rodriguez MG, Ickovics JR. Group prenatal care and improved birth outcomes: Results from a type 1 hybrid effectiveness-implementation study. Prev Med. 2021 Dec;153:106853. doi: 10.1016/j.ypmed.2021.106853. Epub 2021 Oct 20. PMID 34678329
- [Derived] Cunningham SD, Lewis JB, Thomas JL, Grilo SA, Ickovics JR. Expect With Me: development and evaluation design for an innovative model of group prenatal care to improve perinatal outcomes. BMC Pregnancy Childbirth. 2017 May 18;17(1):147. doi: 10.1186/s12884-017-1327-3. PMID 28521785